CLINICAL TRIAL: NCT01927419
Title: Phase 2, Randomized, Double Blinded, Study of Nivolumab (BMS-936558) in Combination With Ipilimumab vs Ipilimumab Alone in Subjects With Previously Untreated, Unresectable or Metastatic Melanoma
Brief Title: Study of Nivolumab (BMS-936558) Plus Ipilimumab Compared With Ipilimumab Alone in the Treatment of Previously Untreated, Unresectable, or Metastatic Melanoma
Acronym: CheckMate 069
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA209-069; 2013-002018-11 (EudraCT Number)
Record Dates: First submitted 2013-08-20; First posted 2013-08-22 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2022-03-18 (Actual); Status verified 2022-02

CONDITIONS: Unresectable Melanoma; Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab + Ipilimumab (Experimental): Participants received (Part 1) 1 mg/kg of nivolumab + 3 mg/kg of ipilimumab solution intravenously every 3 weeks for 4 doses (4 cycles), then (Part 2) 3 mg/kg of nivolumab intravenously every 2 weeks until documented disease progression, toxicity, withdrawal of consent, or study completion.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Placebo + Ipilimumab (Experimental): Participants received (Part 1) placebo-matching nivolumab + 3 mg/kg of ipilimumab solution intravenously every 3 weeks for 4 doses (4 cycles), then (Part 2) placebo-matching nivolumab solution intravenously every 2 weeks until documented disease progression, toxicity, withdrawal of consent, or study completion.
  Interventions: Drug: Ipilimumab; Drug: Placebo

INTERVENTIONS:
Drug: Nivolumab
  Other Names: Opdivo, BMS-936558
  Arms: Nivolumab + Ipilimumab
Drug: Ipilimumab
  Other Names: Yervoy
Drug: Placebo — Matching nivolumab
  Arms: Placebo + Ipilimumab

SUMMARY:
The primary purpose of this study is to compare the objective response rate, as determined by investigators, of Nivolumab combined with Ipilimumab versus Ipilimumab monotherapy in patients with untreated, unresectable, or metastatic melanoma

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Key Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status of 0 or 1
* Histologically confirmed unresectable Stage III or Stage IV melanoma
* No prior systemic anticancer therapy for unresectable or metastatic melanoma. Note that prior adjuvant or neoadjuvant melanoma therapy is permitted if it was completed at least 6 weeks prior to date of first dose, and all related adverse events have either returned to baseline or stabilized
* Tumor tissue obtained in the metastatic setting or from an unresectable site must be provided for biomarker analyses and sent to the central laboratory. Biopsy should be excisional, incisional punch, or core needle. Fine needle aspirates or other cytology samples are insufficient
* Known BRAF V600 mutation status as determined by an FDA-approved test. Patients with either V600 wild-type or V600 mutation-positive melanoma are eligible.

Key Exclusion Criteria:

* Active brain metastases or leptomeningeal metastases. Patients with treated brain metastases are eligible if there is no evidence of progression on magnetic resonance imaging scan for at least 8 weeks after completion of treatment and within 28 days prior to first dose of study drug administration. There must also be no requirement for high doses of systemic corticosteroids that could result in immunosuppression (>10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration
* Ocular melanoma
* Patients with active, known, or suspected autoimmune disease. Those with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2013-08-23 (Actual); Primary Completion 2014-07-24 (Actual); Study Completion 2021-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (21):
- United States (19):
  - San Francisco Oncology Associates, San Francisco, California
  - Orlando Health Inc, Orlando, Florida
  - University Of Louisville Medical Center, Inc., Dba, Louisville, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School Of Medicine, St Louis, Missouri
  - Comprehensive Cancer Centers Of Nevada, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University Of New Mexico Cancer Center, Albuquerque, New Mexico
  - NYU Clinical Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - St. Luke's Hospital, Easton, Pennsylvania
  - GHS Cancer Institute, Greenville, South Carolina
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University Of Wisconsin Paul P Carbone Comprehensive Ca Ctr, Madison, Wisconsin
- France (2):
  - Hopital Larrey, Toulouse
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Long GV, Larkin J, Schadendorf D, Grob JJ, Lao CD, Marquez-Rodas I, Wagstaff J, Lebbe C, Pigozzo J, Robert C, Ascierto PA, Atkinson V, Postow MA, Atkins MB, Sznol M, Callahan MK, Topalian SL, Sosman JA, Kotapati S, Thakkar PK, Ritchings C, Pe Benito M, Re S, Soleymani S, Hodi FS. Pooled Long-Term Outcomes With Nivolumab Plus Ipilimumab or Nivolumab Alone in Patients With Advanced Melanoma. J Clin Oncol. 2025 Mar 10;43(8):938-948. doi: 10.1200/JCO.24.00400. Epub 2024 Nov 6. PMID 39504507
- [Derived] Mantia CM, Werner L, Stwalley B, Ritchings C, Tarhini AA, Atkins MB, McDermott DF, Regan MM. Sensitivity of treatment-free survival to subgroup analyses in patients with advanced melanoma treated with immune checkpoint inhibitors. Melanoma Res. 2022 Feb 1;32(1):35-44. doi: 10.1097/CMR.0000000000000793. PMID 34855329
- [Derived] Hodi FS, Chesney J, Pavlick AC, Robert C, Grossmann KF, McDermott DF, Linette GP, Meyer N, Giguere JK, Agarwala SS, Shaheen M, Ernstoff MS, Minor DR, Salama AK, Taylor MH, Ott PA, Horak C, Gagnier P, Jiang J, Wolchok JD, Postow MA. Combined nivolumab and ipilimumab versus ipilimumab alone in patients with advanced melanoma: 2-year overall survival outcomes in a multicentre, randomised, controlled, phase 2 trial. Lancet Oncol. 2016 Nov;17(11):1558-1568. doi: 10.1016/S1470-2045(16)30366-7. Epub 2016 Sep 9. PMID 27622997
- [Derived] Postow MA, Chesney J, Pavlick AC, Robert C, Grossmann K, McDermott D, Linette GP, Meyer N, Giguere JK, Agarwala SS, Shaheen M, Ernstoff MS, Minor D, Salama AK, Taylor M, Ott PA, Rollin LM, Horak C, Gagnier P, Wolchok JD, Hodi FS. Nivolumab and ipilimumab versus ipilimumab in untreated melanoma. N Engl J Med. 2015 May 21;372(21):2006-17. doi: 10.1056/NEJMoa1414428. Epub 2015 Apr 20. PMID 25891304
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 142 participants were randomized, and 140 participants received treatment.
Groups:
- Nivolumab + Ipilimumab: Participants received 1 mg/kg of nivolumab + 3 mg/kg of ipilimumab solution intravenously every 3 weeks for 4 doses (4 cycles), then 3 mg/kg of nivolumab intravenously every 2 weeks until documented disease progression, toxicity, withdrawal of consent, or study completion.
- Ipilimumab: Participants received placebo-matching nivolumab + 3 mg/kg of ipilimumab solution intravenously every 3 weeks for 4 doses (4 cycles), then placebo-matching nivolumab solution intravenously every 2 weeks until documented disease progression, toxicity, withdrawal of consent, or study completion.
Period: Pre-Treatment Period
Arm/Group | Nivolumab + Ipilimumab | Ipilimumab
Started | 95 | 47
Completed | 94 | 46
Not Completed | 1 | 1
Not completed — Adverse event unrelated to study drug | 0 | 1
Not completed — Participants no longer meeting study criteria | 1 | 0
Period: Treatment Period
Arm/Group | Nivolumab + Ipilimumab | Ipilimumab
Started | 94 | 46
Completed | 0 | 0
Not Completed | 94 | 46
Not completed — Disease progression | 17 | 20
Not completed — Study drug toxicity | 48 | 10
Not completed — Death | 0 | 1
Not completed — Adverse event unrelated to study drug | 6 | 3
Not completed — Participant request to discontinue | 12 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Maximum Clinical Benefit | 6 | 2
Not completed — Other reasons | 3 | 4
Not completed — Not Reported | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab + Ipilimumab | Ipilimumab | Total
Number analyzed (Participants) | 95 | 47 | 142
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (11.0) | 64.5 (10.2) | 63.7 (10.7)
Age, Customized [Count of Participants; unit: Participants]
  Younger than 65 years | 48 | 20 | 68
  65 years and older to younger than 75 years | 35 | 22 | 57
  75 years and older | 12 | 5 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 15 | 47
  Male | 63 | 32 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 82 | 43 | 125
  Unknown or Not Reported | 12 | 4 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 92 | 47 | 139
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) - BRAF Wild-type (WT) Participants
Description: Objective Response Rate is defined as the percentage of participants with a best overall response of Complete Response (CR) or Partial Response (PR), assessed by the investigator by using RECIST 1.1 criteria.
  CR=all target and nontarget lesions have disappeared. Lymph nodes selected must have returned to normal size (<10 mm).
  PR=at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: From 12 weeks after Randomization, assessed every 6 weeks up to Week 49 of study treatment and then every 12 weeks until disease progression (up to approximately 76 months)
Population: All randomized BRAF wild-type participants .
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 73 | 37
Percentage of participants | 60.3 [48.1 to 71.5] | 10.8 [3.0 to 25.4]
Statistical Analysis 1: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority; Fisher Exact; Mean Difference (Final Values) = 49.5, 95% CI 2-sided [31.4 to 61.8] — Difference of ORR; Exact 95% CI for difference in ORR uses Newcombe's method
Statistical Analysis 2: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority; Fisher Exact; Odds Ratio (OR) = 12.52, 95% CI 2-sided [3.79 to 52.55]

2. Secondary Outcome: Progression-Free Survival (PFS) - BRAF Wild-type (WT) Participants
Description: PFS is defined as the time between the date of randomization and the first date of documented progression, as assessed by the investigator, or death due to any cause, whichever occurs first. Participants who died without a reported progression were considered to have progressed on the date of their death. Participants who did not progress or died were censored on the date of their last evaluable tumor assessment.
  PFS values are based on Kaplan-Meier Estimates.
Time Frame: From randomization to progression or death (up to approximately 88 months)
Population: All randomized BRAF wild-type participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 73 | 37
Months | 58.41 [7.23 to NA] — Upper Limit value could not be determined to insufficient number of events. | 4.30 [2.76 to 5.32]
Statistical Analysis 1: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority; Unstratified Cox proportional hazard; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.21 to 0.59] — Nivolumab + Ipilimumab over Ipilimumab

3. Secondary Outcome: Objective Response Rate (ORR) - BRAF Mutant Participants
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All randomized BRAF mutant participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 22 | 10
Percentage of participants | 54.5 [32.2 to 75.6] | 10.0 [0.3 to 44.5]
Statistical Analysis 1: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority; Fisher Exact; Mean Difference (Final Values) = 44.5, 95% CI 2-sided [8.2 to 64.8] — Difference of ORR; Exact 95% CI for difference in ORR uses Newcombe's method
Statistical Analysis 2: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority; Fisher Exact; Odds Ratio (OR) = 10.80, 95% CI 2-sided [1.07 to 511.89]

4. Secondary Outcome: Progression-Free Survival (PFS) - BRAF Mutant Participants
Description: as for outcome 2
Time Frame: From randomization to progression or death (up to approximately 88 months)
Population: All randomized BRAF mutant participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 22 | 10
Months | 8.61 [2.79 to NA] — Upper Limit value could not be determined to insufficient number of events. | 2.73 [0.99 to 5.42]
Statistical Analysis 1: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority; Unstratified Cox proportional hazard; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.14 to 0.97] — Nivolumab + Ipilimumab over Ipilimumab

5. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Overall Quality of Life (QOL) C30 Score
Description: The EORTC QLQ-C30 version 3 is a questionnaire developed to assess the QOL of cancer patients. The questionnaire is a 30-item tool, and it comprises 6 functional subscales (physical functioning, role functioning, cognitive functioning, emotional functioning, social functioning and global quality of life) as well as 9 symptom subscales (fatigue, pain, nausea/vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties).
  Scores for each subscale range from 0 to 100. For the 6 functional subscales, a higher score represents a better level of functioning/health status. For the 9 symptom subscales, a lower score represents a better outcome (low level of symptomatology).
  Scores for the 15 subscales are presented individually.
Time Frame: From Baseline (prior to start of study treatment) to Week 25 after first dose
Population: All randomized participants with available measurements at baseline and week 25
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 22 | 13
Score on a scale
  Physical Functioning | 2.12 (17.625) | 1.03 (9.367)
  Role Functioning | -1.52 (22.950) | 5.13 (21.926)
  Emotional Functioning | 8.33 (10.603) | 10.26 (17.063)
  Cognitive Functioning | -1.52 (15.352) | -2.56 (11.479)
  Social Functioning | 2.27 (22.593) | 0.00 (16.667)
  Global Health Status | 3.79 (11.422) | -0.64 (29.357)
  Fatigue | -3.54 (21.520) | -0.85 (17.836)
  Nausea and Vomiting | -3.03 (12.211) | -2.56 (6.259)
  Pain | -2.27 (12.905) | -8.97 (21.099)
  Dyspnea | -9.09 (23.417) | -7.69 (27.735)
  Insomnia | -12.12 (31.782) | -12.82 (16.879)
  Appetite Loss | -13.64 (30.271) | -2.56 (16.452)
  Constipation | -3.03 (20.339) | 0.00 (13.608)
  Diarrhea | -3.03 (14.213) | 5.13 (12.518)
  Financial Difficulties: number analyzed (Participants) | 22 | 12
  Financial Difficulties | -3.03 (22.792) | -2.78 (22.285)

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from date of first dose to study completion (up to approximately 90 months). Serious Adverse events and other adverse events were assessed from date of first dose to 100 days following date of last dose (up to approximately 86 months).
Description: All treated participants
Arm/Group | Nivolumab + Ipilimumab | Ipilimumab
All-Cause Mortality (participants affected / at risk) | 44/94 | 29/46
Serious Adverse Events (participants affected / at risk) | 69/94 | 27/46
Other Adverse Events (participants affected / at risk) | 90/94 | 45/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Ipilimumab (N=94) | Ipilimumab (N=46)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 3 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Endocrine disorder (Endocrine disorders) | 1 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1
Hypophysitis (Endocrine disorders) | 2 | 1
Hypopituitarism (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Autoimmune colitis (Gastrointestinal disorders) | 3 | 2
Colitis (Gastrointestinal disorders) | 13 | 2
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 5
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Oesophageal pain (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Chills (General disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 6 | 4
Hepatitis (Hepatobiliary disorders) | 3 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 3
Sepsis (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0
Amylase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0
Lipase increased (Investigations) | 2 | 1
Transaminases increased (Investigations) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 8
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Meningoradiculitis (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 2
Spinal cord compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0
Embolism (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Ipilimumab (N=94) | Ipilimumab (N=46)
Anaemia (Blood and lymphatic system disorders) | 24 | 15
Atrial fibrillation (Cardiac disorders) | 6 | 3
Sinus tachycardia (Cardiac disorders) | 4 | 3
Tachycardia (Cardiac disorders) | 5 | 5
Ear pain (Ear and labyrinth disorders) | 5 | 1
Adrenal insufficiency (Endocrine disorders) | 7 | 3
Hypophysitis (Endocrine disorders) | 10 | 2
Hypothyroidism (Endocrine disorders) | 18 | 7
Vision blurred (Eye disorders) | 15 | 0
Abdominal discomfort (Gastrointestinal disorders) | 4 | 3
Abdominal distension (Gastrointestinal disorders) | 9 | 3
Abdominal pain (Gastrointestinal disorders) | 20 | 12
Abdominal pain upper (Gastrointestinal disorders) | 9 | 3
Colitis (Gastrointestinal disorders) | 9 | 4
Constipation (Gastrointestinal disorders) | 32 | 14
Diarrhoea (Gastrointestinal disorders) | 54 | 24
Dry mouth (Gastrointestinal disorders) | 9 | 6
Dyspepsia (Gastrointestinal disorders) | 7 | 3
Flatulence (Gastrointestinal disorders) | 4 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 40 | 25
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 4
Vomiting (Gastrointestinal disorders) | 29 | 11
Asthenia (General disorders) | 17 | 11
Chills (General disorders) | 21 | 8
Fatigue (General disorders) | 57 | 34
Influenza like illness (General disorders) | 5 | 6
Malaise (General disorders) | 2 | 3
Mucosal inflammation (General disorders) | 3 | 5
Non-cardiac chest pain (General disorders) | 5 | 4
Oedema peripheral (General disorders) | 26 | 10
Pain (General disorders) | 14 | 10
Peripheral swelling (General disorders) | 3 | 3
Pyrexia (General disorders) | 32 | 17
Pneumonia (Infections and infestations) | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 7 | 5
Urinary tract infection (Infections and infestations) | 9 | 2
Alanine aminotransferase increased (Investigations) | 30 | 7
Amylase increased (Investigations) | 14 | 3
Aspartate aminotransferase increased (Investigations) | 31 | 7
Blood alkaline phosphatase increased (Investigations) | 13 | 7
Blood bilirubin increased (Investigations) | 12 | 1
Blood creatinine increased (Investigations) | 10 | 4
Blood thyroid stimulating hormone decreased (Investigations) | 7 | 1
Blood thyroid stimulating hormone increased (Investigations) | 8 | 0
Lipase increased (Investigations) | 22 | 6
Platelet count decreased (Investigations) | 5 | 0
Weight decreased (Investigations) | 16 | 2
Weight increased (Investigations) | 5 | 3
Decreased appetite (Metabolism and nutrition disorders) | 26 | 17
Dehydration (Metabolism and nutrition disorders) | 22 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 22 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 12 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 9
Dizziness (Nervous system disorders) | 17 | 5
Dysgeusia (Nervous system disorders) | 6 | 1
Headache (Nervous system disorders) | 35 | 11
Paraesthesia (Nervous system disorders) | 9 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 4
Taste disorder (Nervous system disorders) | 5 | 0
Anxiety (Psychiatric disorders) | 7 | 4
Depression (Psychiatric disorders) | 4 | 4
Insomnia (Psychiatric disorders) | 20 | 11
Pollakiuria (Renal and urinary disorders) | 5 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 20
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 5
Erythema (Skin and subcutaneous tissue disorders) | 10 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 8 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 47 | 17
Rash (Skin and subcutaneous tissue disorders) | 45 | 17
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16 | 8
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 | 4
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 5 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 11 | 4
Flushing (Vascular disorders) | 5 | 1
Hot flush (Vascular disorders) | 1 | 3
Hypertension (Vascular disorders) | 12 | 4
Hypotension (Vascular disorders) | 11 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.